CLINICAL TRIAL: NCT02900794
Title: Comparing Post-Operative Outcomes Between Gold Laser and Micro-Debriders for Functional Endoscopic Sinus Surgery (FESS) in Patients With Chronic Sinusitis
Brief Title: Gold Laser Vs. Micro-Debriders for Functional Endoscopic Sinus Surgery
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No enrollment
Sponsor: Texas Tech University Health Sciences Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: L16-117
Record Dates: First submitted 2016-08-22; First posted 2016-09-14 (Estimated); Last update posted 2019-12-10 (Actual); Status verified 2019-12

CONDITIONS: Sinusitis
MeSH Terms: conditions — Sinusitis | interventions — Lasers, Gas

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Contrast Arm (Microdebridement) (Other): Typical pre-operative intervention including injectable local anesthetic into the inferior and middle turbinates followed by topical anesthetic on soaked cottonoids or pledgets placed in the nasal cavity floor, medial to the middle turbinate, behind the uncinate process will be performed. Using endoscopy, the nasal passage is located. Under endoscopic visualization, the microdebrider will be utilized to perform 1) excision of the concha bullosa, 2) maxillary antrostomy, and 3) submucosal cauterization of the turbinates. Suction/irrigation will be utilized as necessary.
  Interventions: Procedure: Microdebridement
- Treatment Arm (Gold Laser) (Other): Typical pre-operative intervention including injectable local anesthetic into the inferior and middle turbinates followed by topical anesthetic on soaked cottonoids or pledgets placed in the nasal cavity floor, medial to the middle turbinate, behind the uncinate process will be performed. Using endoscopy, the nasal passage is located. Under endoscopic visualization, the Gold Laser will be utilized to perform 1) excision of the concha bullosa, 2) maxillary antrostomy, and 3) submucosal cauterization of the turbinates. Suction/irrigation will be utilized as necessary. If the Investigator determines that the sinus is not sufficiently dilated or cannot be accessed, the need for and the type of additional treatment will be at the discretion of the Investigator.
  Interventions: Device: Gold Laser

INTERVENTIONS:
Device: Gold Laser — Under endoscopic visualization, the Gold Laser will be utilized to perform 1) excision of the concha bullosa, 2) maxillary antrostomy, and 3) submucosal cauterization of the turbinates. Suction/irrigation will be utilized as necessary.
  Arms: Treatment Arm (Gold Laser)
Procedure: Microdebridement — Under endoscopic visualization, the microdebrider will be utilized to perform 1) excision of the concha bullosa, 2) maxillary antrostomy, and 3) submucosal cauterization of the turbinates.
  Arms: Contrast Arm (Microdebridement)

SUMMARY:
Sinusitis is a common medical problem, which significantly decreases patients' quality of life (QOL). Patients may have symptoms such as headaches, sinus pressure, nasal congestion and drainage, decreased sense of smell, and malaise. Surgical therapy for sinusitis attempts to restore the sinus health by directly relieving sinus obstruction. Small telescopes, called endoscopes, are placed through the nostrils into the nasal cavity to enhance visualization, illumination, and magnification of the sinuses and adjacent structures. There are a variety of surgical instruments available to a surgeon for ESS such as stainless steel tools (shavers, microdebriders, or grasping tools) to address sinusitis. Surgical therapy has been shown to improve QOL, decrease medication use and days missed at work for subjects. The use of lasers in treatment of chronic sinus infections is well documented. The LF-40 Gold Laser (Medical Energy, Inc.; Pensacola, FL) has already been approved for clinical use in various procedures including tonsillectomy, adenoidectomy, tracheal stenosis (narrowing), post-intubation granuloma, recurrent respiratory papilloma, and microtia (an underdeveloped ear), and sinus surgery. In this study, the investigators plan to utilize the Gold laser for 1) excision of the concha bullosa, 2) maxillary antrostomy, and 3) submucosal cauterization of the turbinates and compare postoperative outcomes with the use of a microdebrider. These uses are under the approved indication for the LF 40 Gold Laser1, 2, 3. The follow-up times are as follows: 2 weeks postoperatively, 2 months postoperatively, 6 months postoperatively.

DETAILED DESCRIPTION:
Sinusitis is a common medical problem, which significantly decreases patients' quality of life (QOL). Patients may have symptoms such as headaches, sinus pressure, nasal congestion and drainage, decreased sense of smell, and malaise. In the United States annually, 30 million cases of sinusitis are diagnosed with an occurrence of 1 in 8 adults. The direct medical costs are estimated at $2.4 billion per year with indirect costs reaching upwards of $5 billion. Rhinosinusitis is described as the symptomatic inflammation of the paranasal sinuses and nasal cavity. The term rhinosinusitis is preferred because most sinusitis is accompanied by inflammation of the contiguous nasal mucosa. Uncomplicated rhinosinusitis is defined as rhinosinusitis without clinically evident extension of inflammation outside the paranasal sinuses and nasal cavity at the time of diagnosis (e.g. no neurologic, ophthalmologic, or soft tissue involvement). Rhinosinusitis may be classified by duration as acute rhinosinusitis (ARS) (<4 weeks' duration) or as chronic rhinosinusitis (CRS) (>12 weeks), with or without acute exacerbations. This condition can resolve spontaneously, but often requires antibiotics and/or steroids, which is successful in a majority of patients. Sinus surgery is therefore indicated in patients whose symptoms persist despite conservative medical management. A guideline providing evidence-based recommendations for the diagnosis and management of adult sinusitis was developed and revised by a panel of physicians, nurses, and healthcare professionals under the support of the American Academy of Otolaryngology - Head and Neck Surgery.

Surgical therapy for sinusitis attempts to restore the sinus health by directly relieving sinus obstruction. Small telescopes, called endoscopes, are placed through the nostrils into the nasal cavity to enhance visualization, illumination, and magnification of the sinuses and adjacent structures. This "endoscopic sinus surgery" or (ESS) techniques have been developed to treat four types of sinuses (maxillary, frontal, sphenoid, and ethmoid). The variability of involvement of the sinuses vary from patient to patient. There are a variety of surgical instruments available to a surgeon for ESS such as stainless steel tools (shavers, microdebriders, or grasping tools) to address sinusitis. Surgical therapy has been shown to improve QOL, decrease medication use and days missed at work for subjects.

The use of lasers has shown to be beneficial in several otolaryngological procedures. The LF-40 Gold Laser (Medical Energy, Inc.; Pensacola, FL) has already been approved for clinical use in various head and neck surgical procedures including functional endoscopic sinus surgery. With the use of the LF-40 Gold Laser, this study is being performed with the intentions of comparing post-operative outcomes with sinus surgeries performed using a microdebrider.

The purpose of this study will be to determine if post operative outcomes while utilizing the gold laser for performing excision of the concha bullosa, maxillary antrostomy, and submucosal cauterization of the turbinates are significantly improved as compared to use of microdebrider for sinus surgeries. The investigators aim to determine the treatment outcomes 2 weeks, 2 months, and 6 months postoperatively as compared to use of a microdebrider.

ELIGIBILITY:
Inclusion Criteria:

* Study will include subjects age 18 or older with chronic rhinosinusitis as described by the guidelines published in the 2015 Clinical practice guideline (update): adult sinusitis of the American Academy of Otolaryngology - Head & Neck Surgery (AAO-HNS).

  1. Males and females aged 18 or greater
  2. Chronic rhinosinusitis as described by the guidelines published in the 2015 Clinical practice guideline (update): adult sinusitis of the American Academy of Otolaryngology - Head & Neck Surgery (AAO-HNS)

     a. >12 weeks of two or more of the following signs i. mucopurulent drainage (anterior, posterior, or both) ii. nasal obstruction or congestion iii. facial pain/pressure or fullness, or iv. decreased ability to smell b. AND inflammation is documented by one or more of the following findings i. Purulent mucus or edema in the middle meatus or ethmoid region ii. Radiographic imaging showing inflammation of the paranasal sinuses
  3. At least one episode of CRS documented in study investigator's practice with an endoscopic examination with purulent drainage and edema at the time consistent with CRS
  4. Radiographic evidence of sinus inflammation during chronic bacterial rhinosinusitis indicating sinus disease at the ostiomeatal complex.
  5. Willing and able to read and sign informed consent form and remain compliant with the protocol and study procedures
  6. Able to read and understand English
  7. Patients whom are planning to have functional endoscopic sinus surgery.

Exclusion Criteria:

* 1. Diagnosis of Acute Rhinosinusitis or recurrent acute rhinosinusitis

  1. per guidelines published in the 2015 Clinical practice guideline (update): adult sinusitis of the American Academy of Otolaryngology - Head & Neck Surgery (AAO-HNS)

     2. Polyps in nasal cavity or the middle meatus

     3. Prior sinus surgery, not including rhinoplasty or septoplasty

     4. Physician determined need for ethmoidectomy, polypectomy, septoplasty

     5. Patients with known immunodeficiency, ciliary dysfunction, uncontrolled diabetes (defined as most recent HgA1C > 5.7), and/or autoimmune disease

     6. Any clinically significant illness that may interfere with the evaluation of the study

     7. Patients who were involved in other clinical studies 6 months prior to the study initiation

     8. Patients unable to adhere to follow-up schedule or protocol requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2018-07 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Total Chronic Sinusitis Survey (CSS) Score | 2 weeks, 8 weeks, 24 weeks
  Comparison will be made of change in patient-reported quality of life (QOL) as measured by Total CSS score at 2 weeks, 8 weeks, and 24 weeks postoperatively for subjects randomized to micro-debridement versus gold laser.

SECONDARY OUTCOMES:
Rhinosinusitis Disability Index (RSDI) Score | 2 weeks, 8 weeks, 24 weeks
  Comparison will be made of change in patient-reported quality of life (QOL) as measured by rhinosinusitis disability index (RSDI) total, physical, functional, and emotional sub-scores at 2 weeks, 8 weeks, and 24 weeks postoperatively for subjects randomized to microdebridement versus gold laser
Number of Patients Reporting Use of Sinusitis Related Medications Post-Surgically (Medications include: Oral antibiotics, Oral steroids, Topical intranasal steroid sprays, Topical and Nasal Anti-histamines) | 8 weeks, 24 weeks
  Comparison will be made of medication type (name), dosage, frequency, and route of administration at 8 weeks and 24 weeks postoperatively (days of oral antibiotics, oral steroids, topical intranasal steroid sprays, topical and nasal anti-histamines) for subjects randomized to microdebridement versus gold laser.
Days Missed At Work/School | 8 weeks, 24 weeks
  Comparison will be made of missed days at work/school and unscheduled medical care visits due to sinusitis at 8 weeks and 24 weeks postoperatively for subjects randomized to microdebridement versus gold laser.
Number of Sinus Infections | 24 Weeks
  Comparison will be made of patient reported pre-post-enrollment sinus infections and patient-reported sinus infection severity for subjects randomized to microdebridement versus gold laser

CONTACTS AND LOCATIONS:
Overall Officials: Joehassin Cordero, MD, Principal Investigator — TTUHSC
Locations (1):
- Texas Tech University Health Sciences Center, Lubbock, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Gerlinger I, Lujber L, Jarai T, Pytel J. KTP-532 laser-assisted endoscopic nasal sinus surgery. Clin Otolaryngol Allied Sci. 2003 Apr;28(2):67-71. doi: 10.1046/j.1365-2273.2003.00660.x. PMID 12680820
- [Background] Blackwell DL, Lucas JW, Clarke TC. Summary health statistics for U.S. adults: national health interview survey, 2012. Vital Health Stat 10. 2014 Feb;(260):1-161. PMID 24819891
- [Background] Benninger MS, Ferguson BJ, Hadley JA, Hamilos DL, Jacobs M, Kennedy DW, Lanza DC, Marple BF, Osguthorpe JD, Stankiewicz JA, Anon J, Denneny J, Emanuel I, Levine H. Adult chronic rhinosinusitis: definitions, diagnosis, epidemiology, and pathophysiology. Otolaryngol Head Neck Surg. 2003 Sep;129(3 Suppl):S1-32. doi: 10.1016/s0194-5998(03)01397-4. No abstract available. PMID 12958561
- [Background] McCaig LF, Hughes JM. Trends in antimicrobial drug prescribing among office-based physicians in the United States. JAMA. 1995 Jan 18;273(3):214-9. PMID 7807660
- [Background] Snow V, Mottur-Pilson C, Hickner JM; American Academy of Family Physicians; American College of Physicians-American Society of Internal Medicine; Centers for Disease Control; Infectious Diseases Society of America. Principles of appropriate antibiotic use for acute sinusitis in adults. Ann Intern Med. 2001 Mar 20;134(6):495-7. doi: 10.7326/0003-4819-134-6-200103200-00016. No abstract available. PMID 11255527
- [Background] Bhattacharyya N. Chronic rhinosinusitis: is the nose really involved? Am J Rhinol. 2001 May-Jun;15(3):169-73. doi: 10.2500/105065801779954184. PMID 11453503
- [Background] Poetker DM, Litvack JR, Mace JC, Smith TL. Recurrent acute rhinosinusitis: presentation and outcomes of sinus surgery. Am J Rhinol. 2008 May-Jun;22(3):329-33. doi: 10.2500/ajr.2008.22.3177. PMID 18588769
- [Background] Metson R. Holmium:YAG laser endoscopic sinus surgery: a randomized, controlled study. Laryngoscope. 1996 Jan;106(1 Pt 2 Suppl 77):1-18. doi: 10.1097/00005537-199601001-00001. PMID 8538352
- [Background] Lee JC, Lai WS, Ju DT, Chu YH, Yang JM. Diode laser assisted minimal invasive sphenoidotomy for endoscopic transphenoidal pituitary surgery: our technique and results. Lasers Surg Med. 2015 Mar;47(3):239-42. doi: 10.1002/lsm.22340. PMID 25810080
- [Background] Chester AC, Sindwani R. Symptom outcomes in endoscopic sinus surgery: a systematic review of measurement methods. Laryngoscope. 2007 Dec;117(12):2239-43. doi: 10.1097/MLG.0b013e318149224d. PMID 18322425
- [Background] Alobid I, Bernal-Sprekelsen M, Mullol J. Chronic rhinosinusitis and nasal polyps: the role of generic and specific questionnaires on assessing its impact on patient's quality of life. Allergy. 2008 Oct;63(10):1267-79. doi: 10.1111/j.1398-9995.2008.01828.x. PMID 18782106
- [Background] Senior BA, Glaze C, Benninger MS. Use of the Rhinosinusitis Disability Index (RSDI) in rhinologic disease. Am J Rhinol. 2001 Jan-Feb;15(1):15-20. doi: 10.2500/105065801781329428. PMID 11258649
- [Background] Benninger MS, Senior BA. The development of the Rhinosinusitis Disability Index. Arch Otolaryngol Head Neck Surg. 1997 Nov;123(11):1175-9. doi: 10.1001/archotol.1997.01900110025004. PMID 9366696
- [Background] Soler ZM, Hyer JM, Karnezis TT, Schlosser RJ. The Olfactory Cleft Endoscopy Scale correlates with olfactory metrics in patients with chronic rhinosinusitis. Int Forum Allergy Rhinol. 2016 Mar;6(3):293-8. doi: 10.1002/alr.21655. Epub 2015 Dec 31. PMID 26718315
- [Background] Rudmik L, Hopkins C, Peters A, Smith TL, Schlosser RJ, Soler ZM. Patient-reported outcome measures for adult chronic rhinosinusitis: A systematic review and quality assessment. J Allergy Clin Immunol. 2015 Dec;136(6):1532-1540.e2. doi: 10.1016/j.jaci.2015.10.012. PMID 26654198
- [Background] Gliklich RE, Hilinski JM. Longitudinal sensitivity of generic and specific health measures in chronic sinusitis. Qual Life Res. 1995 Feb;4(1):27-32. doi: 10.1007/BF00434380. PMID 7711687
- [Background] Gliklich RE, Metson R. Techniques for outcomes research in chronic sinusitis. Laryngoscope. 1995 Apr;105(4 Pt 1):387-90. doi: 10.1288/00005537-199504000-00010. PMID 7715384
- [Background] Smith TL, Kern R, Palmer JN, Schlosser R, Chandra RK, Chiu AG, Conley D, Mace JC, Fu RF, Stankiewicz J. Medical therapy vs surgery for chronic rhinosinusitis: a prospective, multi-institutional study with 1-year follow-up. Int Forum Allergy Rhinol. 2013 Jan;3(1):4-9. doi: 10.1002/alr.21065. Epub 2012 Jun 26. PMID 22736422
- [Background] Metson RB, Gliklich RE. Clinical outcomes in patients with chronic sinusitis. Laryngoscope. 2000 Mar;110(3 Pt 3):24-8. doi: 10.1097/00005537-200003002-00007. PMID 10718411
- See also: Sinus Surgery [Internet]. Pensacola: Medical Energy Inc.; c2015 [cited 2016 March 24] — http://medicalenergy.com/ent-surgery/
- See also: Winters R, Knight Worley N. Gold Laser Resection of the Concha Bullosa: Description of a New Technique. Otolaryngology. 2012; 2:2. — http://www.omicsonline.org/gold-laser-resection-of-the-concha-bullosa-description-of-a-new-technique-2161-119X.1000114.php?aid=6422
- See also: Lethbridge-Cejku M, Rose D, Vickerie J. Summary health statistics for US adults: National Health Interview Survey, 2004. Vital Health Stat. 2006;10:19-22. — http://www.cdc.gov/nchs/data/series/sr_10/sr10_228.pdf
- See also: Stavem K, Rossberg E, Larsson P. Reliability, validity and responsiveness of a Norwegian Version of the Chronic Sinusitis Survey. BMC Ear, Nose and Throat Disorders. 2006; 6:9. — http://bmcearnosethroatdisord.biomedcentral.com/articles/10.1186/1472-6815-6-9
- See also: 1. Ware, JE. The SF-36 Health Survey Manual and Interpretation Guide. Nimrod Press, Boston 1993; pp 10-14 — http://czresearch.com/info/SF36_healthsurvey_ch6.pdf